CLINICAL TRIAL: NCT01095432
Title: Partial Wave Spectroscopic Detection of Colon Cancer Risk
Acronym: Brushings
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-066-B
Record Dates: First submitted 2010-03-24; First posted 2010-03-30 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis; Colon Cancer
Keywords: Colonoscopy; Flexible Sigmoidoscopy
MeSH Terms: conditions — Colitis, Ulcerative; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of rectal mucosa will be collected during the subject's standard of care colonoscopy or flexible sigmoidoscopy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main Study Group: All subjects who are undergoing a standard of care colonoscopy for flexible sigmoidoscopy and have a history of UC and agree to participate will be in the main study group.
  Interventions: Procedure: PWS Testing

INTERVENTIONS:
Procedure: PWS Testing — Partial wave spectroscopy (PWS)has been developed to allow scientists to learn about any changes to the cells that may indicate a risk of developing colon cancer.

SUMMARY:
The purpose of this study is to study samples of rectal mucosa (the moist lining of the rectum) using a new light scattering technology, called partial wave spectroscopy (PWS) in patients who will undergo a standard of care colonoscopy or a flexible sigmoidoscopy and have a history of ulcerative colitis (UC).

DETAILED DESCRIPTION:
The purpose of this study is to study samples of rectal mucosa (the moist lining of the rectum) using a new light scattering technology, called partial wave spectroscopy (PWS)in patients who will undergo a colonoscopy or a flexible sigmoidoscopy and have a history of ulcerative colitis (UC). PWS has been recently developed to allow scientists to learn about any changes to the cells that may indicate a risk of developing colon cancer. We believe that the PWS test will more accurately detect the risk of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years old or older.
* Patient is already scheduled for a standard of care colonoscopy or flexible sigmoidoscopy.
* Patient has not received chemotherapy.
* History of ulcerative colitis.

Exclusion Criteria:

* Patient is unable to give informed consent..
* Patient has received chemo or radiation therapy within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to undergo a standard of care flexible sigmoidoscopy or a colonoscopy and have a history of UC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Study samples of rectal mucosa (the moist lining of the rectum) using PWS. | 1 year
  Samples will be collected and then shipped to Northwestern University for analysis using PWS. This is to assess accuracy of detecting the risk for colon cancer.

CONTACTS AND LOCATIONS:
Overall Officials: David T Rubin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, DCAM, Chicago, Illinois, United States